CLINICAL TRIAL: NCT06991608
Title: A Non-Interventional Study to Compare Digital Monitoring of Patients With Chronic Spontaneous Urticaria by Telemedicine to Face-to-Face Visits in Germany (DigiMoc)
Brief Title: A Study to Compare Digital Disease Monitoring of Patients With csU (Telemedicine to Face-to-Face Visits) in Germany
Acronym: DigiMoc
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLOU064ADE01
Record Dates: First submitted 2025-05-16; First posted 2025-05-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: NIS
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- arm A: F2F: Monitoring via face to face (F2F) visits
  Interventions: Other: Collection of patient data
- Arm B: Teledermatology: Monitoring via teledermatological visits
  Interventions: Other: Collection of patient data

INTERVENTIONS:
Other: Collection of patient data — This non-interventional study and will not influence treatment decisions

SUMMARY:
This is a multicenter, non-randomized, non-interventional two-cohort study with prospective collection of primary data on monitoring of Chronic spontaneous urticaria (CSU) patients by telemedicine or F2F visits in routine clinical care. This implementation science study will collect data from patients during routine CSU monitoring via F2F visits or teledermatological visits. The study will be representative for the real-world patient CSU population in Germany.

DETAILED DESCRIPTION:
This study will investigate the effect of digital monitoring via teledermatology on patient-reported outcomes (PRO) usage in CSU. The automatic provision of PROs at each digital patient-physician contact will allow simple and time-efficient documentation of current symptoms and might improve patients care.

This study seeks to assess the impact of regular teledermatology-based monitoring on the utilization frequency of PROs in patients with CSU, as compared to the in-person visits F2F. Furthermore, the study aims to gauge the adaption, quality and assessibility of teledermatology of both health care providers and patients .

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above
* Written informed consent for participation obtained from the subject
* Diagnosed chronic spontaneous urticaria
* Medical therapy for CSU
* Concomitant chronic inducible urticaria is allowed
* Willing and be able to perform digital visits

Exclusion Criteria:

• Simultaneous participation in any clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with a physician diagnosis of CSU. Any therapy within the scope of admission will be observed and documented.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Average number of UCT usage per patient | 52 weeks
  Average number of urticaria control test (UCT) usage per patient over the course of 52 weeks will be assessed in the teledermatology arm and in the F2F arm
Total number of contacts per patient | 52 weeks
  Total number of contacts per patient over the course of 52 weeks
Time interval in between visits per patient | 52 weeks
  Time interval in between visits per patient over the course of 52 weeks
Average number of visits in F2F arm | 52 weeks
  Average number of visits in face to face (F2F) arm over the time course of 52 weeks
Average number of contacts in digital arm | 52 weeks
  Average number of contacts in digital arm (stratified for type of contact (video, chat)) over the time course of 52 weeks
Median time of patients in the medical department in F2F arm | 52 weeks
  Median time of a patients in the medical department (time between entry and exit of the office)
Median time of a patient for each digital contact in the digital arm | 52 weeks
  Median time of a patient for each digital contact stratified for type of contact (total time of video call, total time for chat messages)
Score of urticaria control test [UCT] | Baseline, week 52
  UCT is a four-item questionnaire to assess symptom control and quality of life. Each question will be rated from 0 points (no control) to 4 (very well controlled) resulting in a final score from 0 (no disease control) to 16 (complete control)
Score of urticaria activity test 7 [UAS7] | Baseline, week 52
  The UAS7 is a weekly score built up by the sum of hives (wheals; measured via hive severity score [HSS7]) and itch (itch severity score [ISS7]) over one week. For assessment of HSS7, the patient will record the number of wheals twice daily (0 (no hives), 1 (1-6 hives), 2(7-12 hives), 3 (> 12 hives) and the final score is added at the end of the week. To calculate the weekly ISS7, the patient will rate the severity of itch twice daily according to a numeric scale (0 (none) to 3 (severe)). The UAS7 is the sum of the HSS7 score and the ISS7 score. The possible range of the weekly UAS7 score is 0 - 42 (highest activity).
score of dermatology life quality index [DLQI] | Baseline, week 52
  The DLQI is a 10-item general dermatology disability index designed to assess health-related quality of life (HRQoL) in adult subjects with skin diseases such as eczema, psoriasis, acne, and viral warts. Participants rate their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives thinking about the previous 7 days. An overall score is calculated and ranges from 0 to 30 (higher score meaning worse disease related QoL)
Survey to assess satisfaction with current consultations for HCPs and patients | Baseline, week 52
  Participants and their treating HCPs will answer questionnaires assessing their satisfaction with current consultations (retrospectively), as well as satisfaction with the consultation assigned during the study (arm A or arm B). The survey covers questions regarding (digital) disease monitoring and their usefulness/effectiveness in the disease indication of csU, usage of (electronic) PROs and their acceptance in clinical practice, time aspects of the two consultation types, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- Germany (19):
  - Novartis Investigative Site, Hamburg, Hamburg
  - Novartis Investigative Site, Lingen Ems, Lower Saxony
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Ahaus
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Freising
  - Novartis Investigative Site, Gelsenkirchen
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Kamen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Selters

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com